CLINICAL TRIAL: NCT05492942
Title: Records for Alcohol Care Enhancement
Acronym: RACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: H-42631; 4R33AA027597-03 (NIH)
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: Unhealthy alcohol use; Best Practice Advisory (BPA); Clinical care management (CCM); Population health management (PHM); Substance use disorder (SUD)
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — Population Health Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Clinician prompting and Decision Support, Best Practice Advisory (BPA) (No Intervention): Access to an existing BPA for risky alcohol use and alcohol use disorder.
- BPA plus Population Health Management (BPA+PHM) (Experimental): Access to the existing Epic BPA for risky alcohol use and alcohol use disorder + targeted support by a population health manager (PHM).
  Interventions: Behavioral: Best Practice Advisory (BPA) and Population Health Management (PHM)
- BPA plus Clinical Care Management (BPA+CCM) (Experimental): Access to the existing Epic BPA for risky alcohol use and alcohol use disorder + targeted support by a clinician care manager (CCM).
  Interventions: Behavioral: Best Practice Advisory (BPA) and Clinical Care Management (CCM)
- BPA plus Population Health Management plus Clinical Care Management (BPA+PHM+CCM) (Experimental): Access to the existing Epic BPA risky alcohol use and alcohol use disorder + targeted support by a population health manager (PHM) and clinician care manager (CCM)
  Interventions: Behavioral: Best Practice Advisory (BPA) and Population Health Management (PHM) and Clinical Care Management (CCM)

INTERVENTIONS:
Behavioral: Best Practice Advisory (BPA) and Population Health Management (PHM) — A clinician will have continued access to the existing Epic BPA that provides clinical decision support and management for risky alcohol use and alcohol use disorder (AUD). Additionally, a clinician will be supported by a PHM who can access and existing registry of patients with possible or confirmed AUD to examine quality metrics for patients with an AUD on the provider panel. The PHM will circulate quarterly reports to the clinicians in this group to provide performance metric data that indicates the proportion of patients on their primary care panel who are initiating and engaging in AUD treatment. Additionally, the PHM will circulate a weekly report of higher risk patients on the clinician's panel who recently had an acute care visit for AUD and could benefit from outreach for follow-up care. PHM does not directly help clinicians with implementation of care with individual patients, and has no direct patient contact.
  Other Names: BPA+PHM
  Arms: BPA plus Population Health Management (BPA+PHM)
Behavioral: Best Practice Advisory (BPA) and Clinical Care Management (CCM) — A clinician will have continued access to the existing Epic BPA that provides clinical decision support and management for risky alcohol use and alcohol use disorder (AUD). The clinician will be supported by a CCM who will assist in identifying patients who need further assessment on the clinician patient panel. The CCM will conduct outreach to patients regarding alcohol use care, and will communicate with the clinician to help decide potential care plans, and then assist in implementing those plans for patients. The CCM has expertise on how to provide appropriate care to patients and can help patients navigate the complex care system. Further assistance by the CCM may include facilitating prescriptions for clinician sign-off, assuring refills, finding, selecting and coordinating specialty AUD care, and contacting patients to make appointments.
  Other Names: BPA+CCM
  Arms: BPA plus Clinical Care Management (BPA+CCM)
Behavioral: Best Practice Advisory (BPA) and Population Health Management (PHM) and Clinical Care Management (CCM) — A clinician will have continued access to the existing Epic BPA that provides clinical decision support and management for risky alcohol use and alcohol use disorder (AUD). Additionally, a clinician will be supported by a PHM and clinical care manager CCM. The PHM can access and existing registry of patients with possible or confirmed alcohol use disorder to examine quality metrics for patients with an alcohol use disorder on the provider panel. The PHM will circulate quarterly reports to the clinicians in this group to provide summaries of data of those who have initiated or engaged in treatment for alcohol use, as well as a weekly report of higher risk patients on their panel who recently had an acute care visit for AUD and could benefit from outreach for follow-up care. The CCM will assist in identifying patients who need further assessment, and will assist in conducting outreach and implementing care to those patients regarding alcohol use care.
  Other Names: BPA+PHM+CCM
  Arms: BPA plus Population Health Management plus Clinical Care Management (BPA+PHM+CCM)

SUMMARY:
Unhealthy alcohol use (the spectrum from risky consumption through alcohol use disorder, AUD) is a leading cause of preventable death in the US (88,424 deaths annually costing $249 billion a year), and alcohol-related health harms (e.g. AUD itself, cirrhosis) are increasing. Despite high frequency of contacts with the medical system, most people with unhealthy alcohol use do not receive evidence-based interventions due to factors such as stigma, lack of knowledge, challenges with implementing and maintaining tool-based screening, time or prioritization constraints, and more.

Electronic health records (EHRs), Best Practice Advisories (BPA) and registries are known and practical tools to improve management and care of chronic disease by aggregating information about the target population, and by assisting the clinician in reminders, decision support, and disease-specific care management. EHRs may help clinicians identify, assess, treat and monitor care when assisted by targeted staff support such as a clinical care manager (CCM) and population health manager (PHM). These support staff help to track outcomes of care and treatments, allowing for increased engagement with the population, and facilitation of care.

DETAILED DESCRIPTION:
The study team created a live database/registry of patients with unhealthy alcohol use in the Boston Medical Center (BMC) electronic health record (Epic), and updated Epic-based best practice advisories (BPA) and clinical decision support (CDS) (Epic Smart Set) for risky alcohol use and AUD. To improve recognition, management, and overall services provided to patients with AUD, this trial aims to test the impact of these EHR tools (the BPA, CDS, registry and registry-based reporting) for risky alcohol use and AUD by incorporating a population health manager (PHM) and clinical care manager (CCM) to augment reach and support to clinicians, and test the feasibility and effectiveness of leveraging EHRs and targeted supports to improve AUD care. A four-group randomized control trial will be implemented to determine which of four interventions is most effective at increasing rates of initiation and engagement in AUD treatment, as well as other clinical processes and outcomes. The trial will compare the use of the 1) BPA alone (only Epic-based clinician prompting and CDS), 2) BPA + PHM, 3) BPA + CCM, and 4) BPA + PHM + CCM, on the trials' primary, secondary, and exploratory outcomes. Trial results will be assessed by examining outcomes for patients on the clinician's panel.

ELIGIBILITY:
Inclusion Criteria for Clinician Participants:

* Adult (18 years or older)
* Physician or Nurse Practitioner
* Practices Primary Care at Boston Medical Center in the General Internal Medicine (GIM) Primary Care Clinic
* Current position in the practice expected to be unchanged for a minimum of 18 months (not a graduating trainee)

Inclusion Criteria for Patient Participants:

Records (EHR, Medicaid accountable care organizations (ACO) claims) from all patients empaneled (patient is assigned to PCP's primary care panel) by study enrolled clinicians who are:

* Adult (18 years or older)
* Have had at least 1 completed visit in general internal medicine at BMC during the last 18 months.

Exclusion Criteria:

• Clinicians who, at the time of study recruitment, are expected to remain in their BMC GIM position for less than 18 months (e.g. resident or fellow trainees expected to graduate within the study time period).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Hurstak, MD MPH, Principal Investigator — Boston Medical Center, General Internal Medicine
Locations (1):
- General Internal Medicine Primary Care Suites, BU Medical Campus, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Magane KM, Saitz R, Fielman S, LaRochelle MR, Shanahan CW, Pace CA, LaValley M, Penington K, Karzhevsky S, Hurstak E. Supporting primary care clinicians in caring for patients with alcohol use disorder: study protocol for Records for Alcohol Care Enhancement (RACE), a factorial four-arm randomized trial. Addict Sci Clin Pract. 2025 Feb 5;20(1):9. doi: 10.1186/s13722-024-00526-x. PMID 39910606

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only clinicians were consented and enrolled. Randomization and the intervention occurred at the clinician level. Outcomes were observed among primary care patients of randomized clinicians.
Period: Overall Study
Arm/Group | Clinician Prompting and Decision Support, Best Practice Advisory (BPA) | BPA Plus Population Health Management (BPA+PHM) | BPA Plus Clinical Care Management (BPA+CCM) | BPA Plus Population Health Management Plus Clinical Care Management (BPA+PHM+CCM)
Started | 30 | 36 | 34 | 34
12 Months | 28 | 36 | 34 | 33
Completed | 20 | 29 | 26 | 21
Not Completed | 10 | 7 | 8 | 13
Not completed — The clinician did not have an active patient panel eligible for outcome for the full 18 months | 10 | 7 | 8 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinician Prompting and Decision Support, Best Practice Advisory (BPA) | BPA Plus Population Health Management (BPA+PHM) | BPA Plus Clinical Care Management (BPA+CCM) | BPA Plus Population Health Management Plus Clinical Care Management (BPA+PHM+CCM) | Total
Number analyzed (Participants) | 30 | 36 | 34 | 34 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (12) | 34 (11) | 38 (14) | 37 (13) | 37 (12)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 17 | 17 | 27 | 16 | 77
  Male | 13 | 15 | 7 | 18 | 53
  Nonbinary or Missing | 0 | 4 | 0 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 1 | 5 | 13
  Not Hispanic or Latino | 27 | 28 | 33 | 29 | 117
  Unknown or Not Reported | 0 | 4 | 0 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 9 | 12 | 10 | 6 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 1 | 3 | 9
  White | 15 | 15 | 23 | 21 | 74
  More than one race | 1 | 1 | 0 | 1 | 3
  Unknown or Not Reported | 1 | 7 | 0 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percent of New Alcohol Use Disorder (AUD) Diagnosis Episodes That Meet Criteria for AUD Treatment Engagement Among Patients With a New AUD Diagnosis Who Are Empaneled to Randomized Clinicians.
Description: The percent of new AUD diagnosis episodes that meet criteria for AUD treatment engagement among patients with a new AUD diagnosis on a randomized clinician's panel. Engagement is defined as having two or more healthcare services (inclusive of AUD medication) with a diagnosis of AUD within 34 days of meeting initiation, which is defined as having a healthcare service for AUD within 14 days of a new AUD diagnosis. A new AUD diagnosis is defined as a health service in which a patient receives a new AUD diagnosis when there has not been an AUD diagnosis during the prior 194 days, excluding diagnoses assigned in emergency department/detox.
  Outcome is reported at the empaneled patient level.
  Outcome measure time frame is based on definitions of initiation and engagement. Engagement is assessed within 34 days following treatment initiation, and initiation is assessed within 14 days of a new AUD diagnosis (34 days + 14 days =a maximum possible outcome measure time frame of 48 days).
Time Frame: The outcome measure is assessed within 48 days following the date of the new AUD diagnosis, among patients empaneled to randomized clinicians.
Population: The overall number of participants analyzed is randomized clinicians in the study. We have listed the number of randomized clinicians in each study arm. The unit of analysis is new alcohol use disorder diagnoses among patients empaneled to randomized clinicians in each study arm. Data source: Medicaid Claims Data
Measure: Count of Units; unit: New AUD diagnosis episodes
Units Other Than Participants: New AUD diagnosis episodes
Arm/Group | Clinician Prompting and Decision Support, Best Practice Advisory (BPA) | BPA Plus Population Health Management (BPA+PHM) | BPA Plus Clinical Care Management (BPA+CCM) | BPA Plus Population Health Management Plus Clinical Care Management (BPA+PHM+CCM)
Number analyzed (Participants) | 30 | 36 | 34 | 34
Number analyzed (New AUD diagnosis episodes) | 70 | 137 | 97 | 153
New AUD diagnosis episodes | 10 | 11 | 12 | 30

2. Secondary Outcome: Percent of New Alcohol Use Disorder (AUD) Diagnosis Episodes That Meet Criteria for AUD Treatment Initiation Among Patients With a New AUD Diagnosis Who Are Empaneled to Randomized Clinicians
Description: The percent of new AUD diagnosis episodes that meet criteria for AUD treatment initiation among patients with a new AUD diagnosis on a randomized clinician's panel. Initiation is defined as having a healthcare service for AUD within 14 days of a new AUD diagnosis. A new AUD diagnosis is defined as a health service in which a patient receives a new AUD diagnosis when there has not been an AUD diagnosis during the prior 194 days, excluding diagnoses assigned in the emergency department/detox.
  Outcome is reported at the empaneled patient level.
  Outcome measure time frame is based on definitions of initiation. Initiation is assessed within 14 days of a new AUD diagnosis (14 days is the maximum possible outcome measure time frame).
  Outcome is assessed in Medicaid claims.
Time Frame: The outcome measure is assessed within 14 days following the date of the new AUD diagnosis, among patients empaneled to randomized clinicians.
Population: as for outcome 1
Measure: Count of Units; unit: New AUD Diagnosis Episodes
Units Other Than Participants: New AUD Diagnosis Episodes
Arm/Group | Clinician Prompting and Decision Support, Best Practice Advisory (BPA) | BPA Plus Population Health Management (BPA+PHM) | BPA Plus Clinical Care Management (BPA+CCM) | BPA Plus Population Health Management Plus Clinical Care Management (BPA+PHM+CCM)
Number analyzed (Participants) | 30 | 36 | 34 | 34
Number analyzed (New AUD Diagnosis Episodes) | 70 | 137 | 97 | 153
New AUD Diagnosis Episodes | 32 | 38 | 44 | 59

3. Secondary Outcome: Percent of New Alcohol Use Disorder (AUD) Diagnosis Episodes Within Which an AUD Medication is Prescribed Within 90 Days of the New AUD Diagnosis Among Patients Who Are Empaneled to Randomized Clinicians
Description: Percent of new Alcohol Use Disorder (AUD) diagnosis episodes within which an AUD medication is prescribed within 90 days of the new AUD diagnosis among patients who are empaneled to randomized clinicians
  AUD medications include: Naltrexone, Intramuscular (IM) Naltrexone, Acamprosate, or Disulfiram.
  Outcome is reported at the new AUD diagnosis episode level among patients empaneled to randomized clinicians.
  Outcome measure time frame is assessed within 90 days of a new AUD diagnosis.
Time Frame: Outcome measure is assessed 90 days following the date of the new AUD diagnosis, among patients empaneled to randomized clinicians.
Population: The overall number of participants analyzed is randomized clinicians in the study. We have listed the number of randomized clinicians in each study arm. The unit of analysis is new alcohol use disorder (AUD) diagnoses among patients empaneled to randomized clinicians in each study arm. Data Source: Electronic Health Record Data
Measure: Count of Units; unit: New AUD Diagnosis Episodes
Units Other Than Participants: New AUD Diagnosis Episodes
Arm/Group | Clinician Prompting and Decision Support, Best Practice Advisory (BPA) | BPA Plus Population Health Management (BPA+PHM) | BPA Plus Clinical Care Management (BPA+CCM) | BPA Plus Population Health Management Plus Clinical Care Management (BPA+PHM+CCM)
Number analyzed (Participants) | 30 | 36 | 34 | 34
Number analyzed (New AUD Diagnosis Episodes) | 225 | 308 | 312 | 277
New AUD Diagnosis Episodes | 18 | 26 | 28 | 27

4. Secondary Outcome: Number of Boston Medical Center (BMC) Outpatient Encounters With an AUD Billing Diagnosis Within 90 Days of a New AUD Diagnosis, Among Patients Who Are Empaneled to a Randomized Clinician.
Description: Number of Boston Medical Center (BMC) outpatient encounters with an AUD billing diagnosis within 90 days of a new AUD diagnosis, among patients with a new AUD diagnosis who are empaneled to a randomized clinician.
  Outcome is reported at the new AUD diagnosis episode level.
  Outcome measure time frame is assessed within 90 days of a new AUD diagnosis.
Time Frame: The outcome measure is assessed within 90 days following the date of the new AUD diagnosis, among patients empaneled to randomized clinicians.
Population: The overall number of participants analyzed is randomized clinicians in the study. We have listed the number of randomized clinicians in each study arm. The unit of analysis is new alcohol use disorder diagnoses among patients empaneled to randomized clinicians in each study arm. Data Source: Electronic Health Record Data
Measure: Median (Full Range); unit: Number of outpatient AUD encounters
Units Other Than Participants: New AUD Diagnosis Episodes
Arm/Group | Clinician Prompting and Decision Support, Best Practice Advisory (BPA) | BPA Plus Population Health Management (BPA+PHM) | BPA Plus Clinical Care Management (BPA+CCM) | BPA Plus Population Health Management Plus Clinical Care Management (BPA+PHM+CCM)
Number analyzed (Participants) | 30 | 36 | 34 | 34
Number analyzed (New AUD Diagnosis Episodes) | 225 | 308 | 312 | 277
Number of outpatient AUD encounters | 0 [0 to 14] | 0 [0 to 10] | 0 [0 to 12] | 0 [0 to 20]

5. Secondary Outcome: Number of BMC Mental Health Clinician Encounters With an AUD Billing Diagnosis Within 90 Days of a New AUD Diagnosis, Among Patients Who Are Empaneled to a Randomized Clinician.
Description: Number of BMC mental health clinician encounters with an AUD billing diagnosis within 90 days of a new AUD diagnosis, among patients with a new AUD diagnosis who are empaneled to a randomized clinician.
  Outcome is reported at the empaneled patient level.
  Outcome measure time frame is assessed within 90 days of a new AUD diagnosis.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: # AUD visits w/mental health clinician
Units Other Than Participants: New AUD diagnosis episodes
Arm/Group | Clinician Prompting and Decision Support, Best Practice Advisory (BPA) | BPA Plus Population Health Management (BPA+PHM) | BPA Plus Clinical Care Management (BPA+CCM) | BPA Plus Population Health Management Plus Clinical Care Management (BPA+PHM+CCM)
Number analyzed (Participants) | 30 | 36 | 34 | 34
Number analyzed (New AUD diagnosis episodes) | 225 | 308 | 312 | 277
# AUD visits w/mental health clinician | 0 [0 to 4] | 0 [0 to 4] | 0 [0 to 11] | 0 [0 to 11]

6. Secondary Outcome: Number of Referrals for Counseling or Specialty AUD Care Within 90 Days of a New AUD Diagnosis, Among Patients Who Are Empaneled to a Randomized Clinician.
Description: Number of referrals for counseling or specialty AUD care such as the BMC Office Based Addiction Treatment (OBAT), Center for Addiction Treatment for AdoLescent/Young adults who use SubsTances (CATALYST), etc., within 90 days of a new AUD diagnosis, among patients with a new AUD diagnosis who are empaneled to a randomized clinician.
  Outcome is reported at the empaneled patient level.
  Outcome measure time frame is assessed within 90 days of a new AUD diagnosis.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: # of referrals for AUD care
Units Other Than Participants: New AUD Diagnosis Episodes
Arm/Group | Clinician Prompting and Decision Support, Best Practice Advisory (BPA) | BPA Plus Population Health Management (BPA+PHM) | BPA Plus Clinical Care Management (BPA+CCM) | BPA Plus Population Health Management Plus Clinical Care Management (BPA+PHM+CCM)
Number analyzed (Participants) | 30 | 36 | 34 | 34
Number analyzed (New AUD Diagnosis Episodes) | 225 | 308 | 312 | 277
# of referrals for AUD care | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 2] | 0 [0 to 1]

7. Secondary Outcome: Number of BMC AUD Specialty Care Encounters With an AUD Billing Diagnosis Within 90 Days of a New AUD Diagnosis, Among Patients Who Are Empaneled to a Randomized Clinician.
Description: Number of BMC AUD specialty care encounters with an AUD billing diagnosis within 90 days of a new AUD diagnosis, among patients with a new AUD diagnosis who are empaneled to a randomized clinician.
  Outcome is reported at the empaneled patient level.
  Outcome measure time frame is assessed within 90 days of a new AUD diagnosis.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: # of AUD specialty care encounters
Units Other Than Participants: New AUD diagnosis episodes
Arm/Group | Clinician Prompting and Decision Support, Best Practice Advisory (BPA) | BPA Plus Population Health Management (BPA+PHM) | BPA Plus Clinical Care Management (BPA+CCM) | BPA Plus Population Health Management Plus Clinical Care Management (BPA+PHM+CCM)
Number analyzed (Participants) | 30 | 36 | 34 | 34
Number analyzed (New AUD diagnosis episodes) | 225 | 308 | 312 | 277
# of AUD specialty care encounters | 0 [0 to 10] | 0 [0 to 8] | 0 [0 to 4] | 0 [0 to 19]

8. Secondary Outcome: Number of Acute Care Encounters Among Patients With a New AUD Diagnosis Who Are Empaneled to Randomized Clinicians.
Description: Number of acute care encounters (emergency department visits and hospitalizations) within 90 days of a new AUD diagnosis, among patients with a new AUD diagnosis who are empaneled to a randomized clinician.
  Outcome is reported at the empaneled patient level.
  Outcome measure time frame is assessed within 90 days of a new AUD diagnosis.
  Outcome is assessed in Medicaid claims.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Median (Full Range); unit: # of acute care utilization encounters
Units Other Than Participants: New AUD diagnosis episodes
Arm/Group | Clinician Prompting and Decision Support, Best Practice Advisory (BPA) | BPA Plus Population Health Management (BPA+PHM) | BPA Plus Clinical Care Management (BPA+CCM) | BPA Plus Population Health Management Plus Clinical Care Management (BPA+PHM+CCM)
Number analyzed (Participants) | 30 | 36 | 34 | 34
Number analyzed (New AUD diagnosis episodes) | 70 | 137 | 97 | 153
# of acute care utilization encounters | 1 [0 to 22] | 1 [0 to 25] | 2 [0 to 26] | 3 [0 to 20]

9. Secondary Outcome: Number of Acute Care Utilization Encounters With an Alcohol-related Diagnosis Among Patients With a New AUD Diagnosis Who Are Empaneled to Randomized Clinicians
Description: Number of acute care utilization encounters (emergency department visits and hospitalizations), with an alcohol-related diagnosis within 90 days of a new AUD diagnosis, among patients with a new AUD diagnosis on are empaneled to a randomized clinician.
  Outcome is reported at the empaneled patient level.
  Outcome measure time frame is assessed within 90 days of a new AUD diagnosis.
  Outcome is assessed in Medicaid claims.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: # acute care utilization AUD encounters
Units Other Than Participants: New AUD diagnosis episodes
Arm/Group | Clinician Prompting and Decision Support, Best Practice Advisory (BPA) | BPA Plus Population Health Management (BPA+PHM) | BPA Plus Clinical Care Management (BPA+CCM) | BPA Plus Population Health Management Plus Clinical Care Management (BPA+PHM+CCM)
Number analyzed (Participants) | 30 | 36 | 34 | 34
Number analyzed (New AUD diagnosis episodes) | 70 | 137 | 97 | 153
# acute care utilization AUD encounters | 0 [0 to 8] | 0 [0 to 10] | 1 [0 to 8] | 2 [0 to 9]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Clinician Prompting and Decision Support, Best Practice Advisory (BPA) | BPA Plus Population Health Management (BPA+PHM) | BPA Plus Clinical Care Management (BPA+CCM) | BPA Plus Population Health Management Plus Clinical Care Management (BPA+PHM+CCM)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/36 | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/36 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/30 | 0/36 | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT05492942/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT05492942/ICF_000.pdf